CLINICAL TRIAL: NCT03048227
Title: Assessement of the Influence of Continuous Glucose Measurement on Glucose Control of Type 1 Diabetic Patients Treated by Implanted Insulin Pump
Brief Title: Can Continuous Glucose Measurements Help Diabetic Patients Treated With an Implantated Pump?
Acronym: CGMIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: CGM Navigator isn't longer available (October 11, 2019)
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UF9773
Record Dates: First submitted 2017-01-23; First posted 2017-02-09 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Type1diabetes
Keywords: TIDM; Type1diabetes; Implantable Pump; CGM

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Glucose Measurement (CGM) (Experimental): Patients will manage their diabetes with the help of Continuous Glucose Measurements (Abbott Freestyle Navigator II).
  Interventions: Device: Continuous Glucose Measurement (CGM)
- Control (No Intervention): Patients will manage their diabetes as usual as recommended by their care team.

INTERVENTIONS:
Device: Continuous Glucose Measurement (CGM) — Patients will manage their diabetes with the help of Continuous Glucose Measurements (Abbott Freestyle Navigator II).
  Arms: Continuous Glucose Measurement (CGM)

SUMMARY:
During this study, we propose to assess the utility of Continuous Glucose Measurements (CGM) in a group of Type 1 diabetic patients treated with an implanted insulin pump. Patients will participate in two period of 3 months separated by a 3 months washout. During one period, they will use CGM to adapt their insulin therapy while during the other period, they will manage their diabetes with their usual capillary blood glucose meter. We except to observe an increase of time spent in glucose safe range when using CGM.

DETAILED DESCRIPTION:
Glucose control and quality of life of patients with type 1 diabetes with high glucose variability can be improve with use of an implanted pump which delivers insulin by the intra-peritoneal route. Some patients however still have difficulties to achieve their glycemic goal despite this therapy. Continuous Glucose Measurements (CGM) has proven to be able to improve glucose control (HbA1c, time spent in hypoglycaemia) of patients treated with an external insulin pump. No trial has been performed yet to assess the utility of CGM on patients using an intra-peritoneal insulin delivery.

During this study, we propose to assess the influence of CGM use on type 1 diabetic subject treated with implanted insulin pump. It is a prospective, randomized cross-over study. After a 2 weeks run-in period with CGM followed by a 4 weeks break, subjects will participate at two experimental periods of 3 months separated with a 3 month washout. During the intervention phase, patient will use a CGM system (Abbott Freestyle Navigator II) to adapt their insulinotherapy. During the control period, patients will based their insulinotherapy upon their usual care and capillary glucose measurements. The order of the periods will be randomized.

The main endpoint will be the time spent in glucose interval 70-180mg/dL during the last 20 days of each period. The control arm will wear a blinded sensor during this phase to allow comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 and 70
* Type 1 diabetes for at least 1 year
* Treatment of diabetes withimplanted insulin pump for at least 6 months
* HbA1c level between 7.5 and 10%
* Minimum of 4 capillary glucose controls per day over past 3 months
* Use of CGM at least 75% during run-in period
* Willingness to follow all study procedures
* Informed consent signed
* Patient must be affiliated or beneficiary of a social medical insurance

Exclusion Criteria:

* Pregnancy of breast feeding, or intention to be pregnant during the study duration
* Impaired cognitive or psychological abilities which may result in defective adherence to study procedures
* Any disease which could make the use glucose sensor difficult (ex : blindness, severe arthrosis or immobility)
* Known allergy to medical adhesive or glucose sensor component
* Medication affecting glucose metabolism, unless stable during the study
* Long term use of continuous glucose measurements during pas 6 months
* Pump implanted more than 6 years ago
* Anti-insulin antobodies syndrom
* Active enrollment in another clinical trial or participation in a study within 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Time spent with glucose | last 20 days of intervention period
  Time spent with glucose between 70-180mg/dL

SECONDARY OUTCOMES:
HbA1c | last 20 days of intervention period
  HbA1c
Time spent in hypoglycaemia | last 20 days of intervention period
  Time spent in hypoglycaemia (<70mg/dL)
Time spent in hyperglycemia | last 20 days of intervention period
  Time spent in hyperglycemia (>180mg/dL)
Time spent in glucose range | last 20 days of intervention period
  Time spent in glucose range [70-180] and [80-140] mg/dL
Glucose mean and standard deviation | last 20 days of intervention period
  Glucose mean and standard deviation
Low Blood Glucose Index (LBGI) | last 20 days of intervention period
  Low Blood Glucose Index (LBGI)
High Blood Glucose Index (HBGI) | last 20 days of intervention period
  High Blood Glucose Index (HBGI)
Glucose Variability | last 20 days of intervention period
  Glucose Variability: MARD : Mean Absolute Relative Difference
Glucose Variability | last 20 days of intervention period
  Glucose Variability: MAGE : Mean Amplitude of Glucose Excursions
  -MODD : Mean Of daily blood Glucose Difference
Glucose Variability | last 20 days of intervention period
  Glucose Variability: MODD : Mean Of daily blood Glucose Difference
Number of symptomatique hypoglycaemia, severe et non severe | last 20 days of intervention period
  Number of symptomatique hypoglycaemia, severe et non severe
Number of pump programmation | last 20 days of intervention period
  Number of pump programmation
Percentage of sensor use | last 20 days of intervention period
  Percentage of sensor use
Score of Quality of Life questionnaire (IDSRQ) | last 20 days of intervention period
  Score of Quality of Life questionnaire (IDSRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Eric RENARD, MD, Principal Investigator — University Hospital, Montpellier
Locations (10):
- France (10):
  - Chu de Nancy, Nancy, Vandoeuvre-les-nancy
  - CHU de Bordeaux, Bordeaux
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU de Dijon, Dijon
  - CHRU de Lille, Lille
  - AP - Hôpitaux de Marseille, Marseille
  - UHMontpellier, Montpellier
  - AP - Hôpitaux de Paris, Paris
  - CHRU de Strasbourg, Strasbourg
  - Chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided
NC